CLINICAL TRIAL: NCT04370288
Title: The Clinical Trial of Application of Methylene Blue Vial for Treatment of Covid-19 Patients
Brief Title: Clinical Application of Methylene Blue for Treatment of Covid-19 Patients
Acronym: Covid-19
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Daryoush Hamidi Alamdari, Associate professor, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IR.MUMS.REC.1399.122
Record Dates: First submitted 2020-04-29; First posted 2020-04-30 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Covid-19
Keywords: Covid-19; Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Methylene Blue; Ascorbic Acid; Acetylcysteine; hydromethylthionine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Covid-19 patients treated with standard medical therapy (supportive therapy).
- Intervention group (Experimental): Covid-19 patients treated with mixture of MCN (Methylene blue, vitamin C, N-acetyl cysteine).
  Interventions: Drug: MCN (Methylene blue, vitamin C, N-acetyl cysteine)

INTERVENTIONS:
Drug: MCN (Methylene blue, vitamin C, N-acetyl cysteine) — A mixture of MCN will be injected to covid-19 patients.
  Other Names: Leucomethylene Blue
  Arms: Intervention group

SUMMARY:
The severe acute respiratory syndrome caused by COVID-19 is now a global catastrophic event. Currently there is no approved drug or vaccine for the disease. Methylene blue (MB, oxidized form, blue color) has been used in many different areas of clinical medicine, ranging from malaria to orthopedics. Leucomethylene Blue (reduced form of MB, colorless) may be applied for the treatment of COVID-19 according to the scientific evidences.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed case of Covid-19 (by RT-PCR, HRCT)
2. Admission to Intensive Care Unit
3. Need for intubation and mechanical ventilation (PaO2/FiO2 < 100-200)
4. Written informed consent

Exclusion Criteria:

1. Pregnancy and breastfeeding
2. History of G6PDH deficiency
3. Preadmission anticoagulation
4. Severe renal insufficiency (glomerular filtration rate <30 mL/min/1.73m2)
5. Medical records of cirrhosis
6. Active chronic hepatitis
7. Severe hepatic disease defined by GOT or GPT levels three times above the normal upper limit
8. Patients with history of allergic reaction or significant sensitivity to Methylene blue
9. Treatment with immunosuppressive agents
10. Use of other investigational drugs in the moment of inclusion

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-04-19 (Actual); Primary Completion 2020-09-20 (Estimated); Study Completion 2020-09-21 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients remaining free of need for mechanical ventilation in both groups | Day 7
  All patient will be assess for changes in disease severity.

SECONDARY OUTCOMES:
Mortality rate in both groups | Day 28
Improvement in Pa02/Fi02 ratio in both groups | Day 2
Duration of hospital stay in both group. | Day 28
Duration of Intensive Care Unit stay in both groups | Day 28
Days free of dialysis in both groups | Day 28
C-reactive proteins | 3-5 Days
WBC Count | 3-5 Days

CONTACTS AND LOCATIONS:
Overall Officials: Daryoush Hamidi Alamdari, Ph.D, Principal Investigator — Mashhad University of Medical Sciences, Mashhad, Iran
Locations (1):
- Imam Reza Hospital, Mashhad, Razavi Khorasan Province, Iran

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- [Derived] Hamidi-Alamdari D, Hafizi-Lotfabadi S, Bagheri-Moghaddam A, Safari H, Mozdourian M, Javidarabshahi Z, Peivandi-Yazdi A, Ali-Zeraati A, Sedaghat A, Poursadegh F, Barazandeh-Ahmadabadi F, Agheli-Rad M, Tavousi SM, Vojouhi S, Amini S, Amini M, Majid-Hosseini S, Tavanaee-Sani A, Ghiabi A, Nabavi-Mahalli S, Morovatdar N, Rajabi O, Koliakos G. METHYLENE BLUE FOR TREATMENT OF HOSPITALIZED COVID-19 PATIENTS: A RANDOMIZED, CONTROLLED, OPEN-LABEL CLINICAL TRIAL, PHASE 2. Rev Invest Clin. 2021;73(3):190-198. doi: 10.24875/RIC.21000028. PMID 34019535
- [Derived] Alamdari DH, Moghaddam AB, Amini S, Keramati MR, Zarmehri AM, Alamdari AH, Damsaz M, Banpour H, Yarahmadi A, Koliakos G. Application of methylene blue -vitamin C -N-acetyl cysteine for treatment of critically ill COVID-19 patients, report of a phase-I clinical trial. Eur J Pharmacol. 2020 Oct 15;885:173494. doi: 10.1016/j.ejphar.2020.173494. Epub 2020 Aug 20. PMID 32828741